CLINICAL TRIAL: NCT00526695
Title: Effects of Sevoflurane in Subanesthetic Concentrations on the Forearm Perfusion, Leukocyte/Thrombocyte Activation, and Endothelial Function After Tourniquet-Induced Ischemia/Reperfusion Injury in the Forearm of Volunteers
Brief Title: Effects of Sevoflurane in Subanesthetic Concentrations on the Forearm Perfusion
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Michael Zaugg, Anesthesiology, Univ. Hospital Zurich
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 17-2005
Record Dates: First submitted 2007-08-27; First posted 2007-09-10 (Estimated); Last update posted 2008-07-18 (Estimated); Status verified 2008-07

CONDITIONS: Ischemia/Reperfusion Injury
Keywords: Ischemia/Reperfusion; Organ Protection; Anesthetics
MeSH Terms: conditions — Reperfusion Injury; Ischemia | interventions — Sevoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sevoflurane (Preconditioning) — Inhalation of sub-anesthetic doses of sevoflurane

SUMMARY:
Sevoflurane preconditioning and cardiovascular protection against ischemia/reperfusion injury.

Study hypothesis: The volatile anesthetic sevoflurane at subanesthetic concentrations achieves endothelial protection against ischemia/reperfusion injury and reduces inflammatory markers in the circulation

DETAILED DESCRIPTION:
Healthy volunteers are included in the study to investigate endothelial function and platelet activation after preconditioning by sevoflurane in subanesthetic concentrations.

Forearm perfusion, endothelial function and leukocyte/thrombocyte activation after tourniquet-induced ischemia/reperfusion injury of the forearm are measured using healthy volunteers in a cross-over design.

ELIGIBILITY:
Inclusion criteria: male

* Non-smoker
* No asthma
* NPO
* Volunteer

Exclusion criteria:

* Female
* Chronic medication
* Asthma
* Smoking

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2005-01; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
marker expression on blood cells | December 2008

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zaugg, PD Dr. med., Principal Investigator — UniversitaetsSpital Zuerich; Michael Zaugg, PD Dr. med., Principal Investigator — University of Zurich
Locations (1):
- University Hospital of Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Lucchinetti E, Zeisberger SM, Baruscotti I, Wacker J, Feng J, Zaugg K, Dubey R, Zisch AH, Zaugg M. Stem cell-like human endothelial progenitors show enhanced colony-forming capacity after brief sevoflurane exposure: preconditioning of angiogenic cells by volatile anesthetics. Anesth Analg. 2009 Oct;109(4):1117-26. doi: 10.1213/ANE.0b013e3181b5a277. PMID 19762739